CLINICAL TRIAL: NCT04125667
Title: Culture System for Isolating Circulating Tumor Cells
Brief Title: Culture System for Isolating Circulating Tumor cells_2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019071239RINB
Record Dates: First submitted 2019-10-02; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-09

CONDITIONS: Early Diagnosis; Diagnostic Techniques and Procedures
Keywords: Circulating cancer cells; Biomedical polymer material; Cell affinity difference; White blood cell attachment
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This culture system utilizes the special affinity difference of biomedical material coating for different cells to achieve the effect of isolating tumor cells from the blood sample. The coating of the system has the characteristic that to make the WBCs adhesion, but the cancer cells in the blood sample suspend in the culture medium, which achieves the effect of separating cancer cells from the blood. The supernatant with the cancer cells can further be isolated from the cultural system for related analysis and detection to achieve early diagnosis and screening.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lung cancer are between the ages of 20 and 70
* Willing to sign the consent form under the informed consent

Exclusion Criteria:

* Vulnerable Subjects included minors, prisoners, aborigines, pregnant women, people with mental disorders, students, and subordinates, etc.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all stages of lung cancer patients between the ages of 20 and 70. Also, to protect the vulnerable subjects, we don't recruit minors, prisoners, aborigines, pregnant women, people with mental disorders, students, and subordinates, etc.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-10-31 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
The Number of Circulating Cancer Cells from The Blood Sample | about 1 week
  The number of circulating cancer cells from the blood sample will be investigated. To distinguish cancer cells from blood cells for the system, the lung cancer cells were immunofluorescence stained for Cytokeratin, white blood cells were stained for CD45 and nuclei were counterstained with DAPI.

SECONDARY OUTCOMES:
Cancer Cell Isolation Efficiency of The Isolation System | about 1 week
  The cell isolation efficiency was characterized by spiking A549 lung cancer cells with celltracker at the concentrations 1000, 100 and 10 cells into whole blood.

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Horng Young, Study Chair — Institute of Biomedical Engineering, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan